CLINICAL TRIAL: NCT03636074
Title: Effects of Hypothermia on Delayed Neurocognitive Recovery: an Observational Trial Among Patients Undergoing Cardiac-Surgery
Brief Title: Effects of Hypothermia on Delayed Neurocognitive Recovery (DNR): an Observational Trial Among Patients Undergoing Cardiac-Surgery
Acronym: DNR
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal Investigator, University of Padova
Other Study IDs: Zivago
Record Dates: First submitted 2018-08-07; First posted 2018-08-17 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Cognitive Dysfunction; Emergence Delirium; Hypothermia
MeSH Terms: conditions — Cognitive Dysfunction; Emergence Delirium; Hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hearth-valve surgery
  Interventions: Procedure: Hypothermia during Extracorporeal Circulation
- Hearth bypass surgery
  Interventions: Procedure: Hypothermia during Extracorporeal Circulation

INTERVENTIONS:
Procedure: Hypothermia during Extracorporeal Circulation — Normothermia during Extracorporeal Circulation

SUMMARY:
Post-operative cognitive dysfunction is a common disease in patient undergoing general anaesthesia, especially in older patients. No correlations have been yet studied between intraoperative hypothermia and incidence of Delayed Neurocognitive Recovery. Investigators are going to estimate the Relative Risk of Hypothermia and emergence of Post-operative cognitive dysfunction in cardiac-surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing Cardiac - Surgery intervention with extracorporeal circulation

Exclusion Criteria:

* Neurological disease before surgery
* Sedation in Cardiac-Surgery Intensive Unit > 6 hours
* Cerebral regional Oxygen saturation <20% baseline during surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective Observational Case-Control
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Delayed Neurocognitive Recovery in Cardiac-Surgery | Patients will be subjected to Montreal Cognitive Assessment and Short Portable Mental Status Questionnaire test one day before surgery and 4-6 days after surgery
  Discover changes between pre-operative general cognition tests (Montreal Cognitive Assessment and Short Portable Mental Status Questionnaire) test score and post-operative Montreal Cognitive Assessment test score.
Incidence of Delayed Neurocognitive Recovery in Cardiac-Surgery | Patients will be subjected to Trail Making Test A and B one day before surgery and 4-6 days after surgery
  Discover changes between pre-operative Trail Making Test A and B score and post-operative Trail Making Test A and B score.
Incidence of Delayed Neurocognitive Recovery in Cardiac-Surgery | Patients will be subjected to Digit Span Test one day before surgery and 4-6 days after surgery
  Discover changes between pre-operative Digit Span Test score and post-operative Digit Span Test score.
Incidence of Delayed Neurocognitive Recovery in Cardiac-Surgery | Patients will be subjected to Frontal Assessment Battery test one day before surgery and 4-6 days after surgery
  Discover changes between pre-operative Frontal Assessment Battery test score and post-operative Frontal Assessment Battery test score and

SECONDARY OUTCOMES:
Effects of hypothermia during Extracorporeal Circulation in Cardiac Surgery | One day before surgery and 4-6 days after surgery patients will be subjected to cognitive test to diagnosticate Post-Operative Cognitive Decline
  Discover statistical significance difference in incidence of Post-Operative Cognitive Decline between patients undergoing normothermia and patients undergoing hypothermia during Extracorporeal Circulation in Cardiac Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided